CLINICAL TRIAL: NCT01402791
Title: Endometriosis: Sexual Dysfunction and Adaptation Strategies Among Couples
Acronym: DYSEXTRIOSE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2011/SD-05; 2011-A00564-37 (Other: RCB number)
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: All patients included according to state inclusion and exclusion criteria.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — All included couples (women and their partners) are required to fill out several questionnaires: 1. Questionnaire for women; 2. Self-questionnaire for women; 3. SFQ for women; 4. Questionnaire for men; 5. Self-questionnaire for men; 6. IIEF for men.

SUMMARY:
The primary objective of this study is to evaluate the presence/absence and description of persistent sexual troubles following surgical treatment for endometriosis for women, and their partners.

ELIGIBILITY:
Inclusion Criteria:

* The patient (and her partner) must have given his/her informed and signed consent
* The patient (and her partner) must be insured or beneficiary of a health insurance plan
* Couples for whom the woman has formerly undergone surgical treatment for endometriosis, and for the partner agrees to respond to questionnaires for this study

Exclusion Criteria:

* The patient (or her partner) is participating in another study
* The patient (or her partner) is in an exclusion period determined by a previous study
* The patient (or her partner) is under judicial protection, under tutorship or curatorship
* The patient (or her partner) refuses to sign the consent
* It is impossible to correctly inform the patient (or her partner)
* The patient is pregnant
* The patient is breastfeeding
* The patient was surgically treated for endometriosis, but was single.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Couples for whom the women have been surgically treated for deep endometriosis at the Nîmes University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Score for the SFQ questionnaire | Day 1
  Score for the SFQ questionnaire; varies from 0 to 5.
Score for the IIEF questionnaire | Day 1
  Score for the IIEF questionnaire; varies from 0 to 75.

SECONDARY OUTCOMES:
Scores for each sub-domain of the SFQ questionnaire | Day 1
  Scores for each sub-domain of the SFQ questionnaire; varies from 0 to 5.
Scores for each sub-domain of the IIEF questionnaire | Day 1
  Scores for each sub-domain of the IIEF questionnaire; varies from 0 to 30.
Sexual treatment request (yes/no) | Day 1
  Did the patients request treatment/help for sexual problems? yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Droupy, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France